CLINICAL TRIAL: NCT03111420
Title: Pivotal Study of the AggreGuide A-100 Adenosine Diphosphate (ADP) Assay to Evaluate the Detection of Platelet Dysfunction Due to P2Y12 Antiplatelet Drugs
Brief Title: Study of AggreGuide A-100 (ADP) Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aggredyne, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: VAL-0085
Record Dates: First submitted 2017-04-02; First posted 2017-04-12 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-05

CONDITIONS: Risk Factor, Cardiovascular; Platelet Dysfunction Due to Drugs
MeSH Terms: interventions — Clopidogrel; Prasugrel Hydrochloride; Ticagrelor; Platelet Function Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Platelet function test results are not provided to the participant, care provider, or investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Clopidogrel (Experimental): Platelet function test before and after administration of P2Y12 inhibitor antiplatelet therapy after ASA 81 mg.
  Loading dose day 1. Maintenance dose over subsequent 7 days.
  Interventions: Drug: P2Y12 inhibitor; Device: Platelet function test
- Prasugrel (Experimental): Platelet function test before and after administration of P2Y12 inhibitor antiplatelet therapy after ASA 81 mg.
  Loading dose day 1. Maintenance dose over subsequent 7 days.
  Interventions: Drug: P2Y12 inhibitor; Device: Platelet function test
- Ticagrelor (Experimental): Platelet function test before and after administration of P2Y12 inhibitor antiplatelet therapy after ASA 81 mg.
  Loading dose day 1. Maintenance dose over subsequent 7 days.
  Interventions: Drug: P2Y12 inhibitor; Device: Platelet function test

INTERVENTIONS:
Drug: P2Y12 inhibitor — Administration of P2Y12 inhibitor antiplatelet therapy
  Other Names: clopidogrel; prasugrel; ticagrelor
Device: Platelet function test — Blood is drawn for testing of platelet aggregation activity
  Other Names: AggreGuide A-100 ADP assay

SUMMARY:
Study to evaluate the performance of the AggreGuide A-100 ADP assay for detection of platelet dysfunction caused by P2Y12 inhibitor antiplatelet therapy.

DETAILED DESCRIPTION:
Study subjects will have A-100 ADP measurements performed at baseline and after initiation of P2Y12 inhibitor antiplatelet therapy, following loading and maintenance doses.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a history of cardiovascular disease OR
* Subject has 2 or more cardiac risk factors:

  * Smoking
  * Hypertension
  * Hyperlipidemia
  * Family History of Heart Disease
  * Post-menopausal female
  * Diabetes
  * Obesity (BMI > 30)
  * Sedentary lifestyle

Exclusion Criteria:

Taken nonsteroidal anti-inflammatory drugs (NSAIDs) drugs, anti-platelet drugs or anticoagulant drugs within the past seven (7) days, over age 75, under 60 kg body weight, in the last trimester of pregnancy or breastfeeding, with a diagnosed history of: stroke or transient ischemic attacks, or other thromboembolic disease, anemia, thrombocytopenia, uncontrolled hypertension,platelet disorders,hemophilia or other bleeding disorder, gastrointestinal disease, severe renal disease, expect to engage in contact sports, scheduled for elective surgery, have a medical history as determined by the Investigator that would pose safety concerns, or possess contraindications for any of the study medications.

Ages: 22 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in Platelet Activity Index (PAI) | Baseline, day 1, day 7
  Platelet reactivity measurement using A-100 ADP assay

CONTACTS AND LOCATIONS:
Overall Officials: Phil Speros, Study Director — Aggredyne, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurbel PA, Tantry US, Bliden KP, Fisher R, Sukavaneshvar S, Dahlen J, Speros PC. Clinical validation of AggreGuide A-100 ADP, a novel assay for assessing the antiplatelet effect of oral P2Y12 antagonists. J Thromb Thrombolysis. 2021 Jul;52(1):272-280. doi: 10.1007/s11239-021-02498-0. Epub 2021 Jun 18. PMID 34143384